CLINICAL TRIAL: NCT07136090
Title: OMERACT Systemic Lupus Erythematosus Delphi Survey Via REDCap
Brief Title: OMERACT SLE Delphi
Status: Not yet recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: OMERACT (Unknown)
Responsible Party: Principal Investigator, Zahi Touma, Principal Investigator, University Health Network, Toronto
Other Study IDs: 24-5926
Record Dates: First submitted 2025-07-09; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: SLE - Systemic Lupus Erythematosus
Keywords: Core Outcome Set
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient cohort: Those with lived experience of systemic lupus erythematosus
- Other Stakeholder cohort: Clinicians, researchers, payors, policy makers, pharmaceutical industry, regulators

SUMMARY:
SLE is a chronic multi-systemic autoimmune disease with clinical manifestations characterized by recurrent flares in disease activity and damage in several organs. SLE affects primarily women during child bearing age and is negatively related to productivity, social role participation and health-related quality of life. The multi-systemic nature of SLE and its diverse clinical manifestations have led to many outcome measurements being utilized in SLE clinical trials and longitudinal studies. To standardize measurement in clinical trials and longitudinal studies, the OMERACT SLE Group developed the core domain set for SLE in 1998. A core domain set is a set of outcome measures, capturing all the facets/aspects of the disease, that standardizes measurement and research across clinical trials and longitudinal studies necessary for the advancement of the field. Since development in 1998, many new important domains for SLE have been identified, thus there is an unmet need to update the core domain set. A new OMERACT SLE Working Group has been established to update the SLE core domain set.

This is a qualitative study that aims to prioritize domains to include in the SLE core domain set. All participants will be asked to complete a four-round online survey. During rounds 1-3 participants will be asked to rate the importance of each domain to be included; round 4 will ask participants select and rank domains. Participants will also have the option of adding other items or descriptors and to provide any other feedback. Each round of the survey will take approximately 15-20 minutes to complete.

Participants will need to participate in round 1 in order to be invited to round 2, and then participate in round 2 in order to be invited to round 3, and final participate in round 3 in order to be invited to round 4.

DETAILED DESCRIPTION:
Objective Research question • What domains (outcome measurements) of SLE are important to the various SLE stakeholders?

Objective

• The investigators are attempting to ascertain preliminary opinions on the importance of domains measured in SLE.

Study Design Constructing e-Delphi Survey Domains REDCap will be used to assist the working group in prioritizing domains for a Core Domain Set and providing decision-making information. The investigators qualitative work and literature reviews have generated 25 domains for consideration across all Core Areas. Based on the investigator's previous qualitative work and literature review, brief definitions have been created for each domain to clarify its meaning. The domains, the core area they represent, and their definitions are included in are included in the accompanying Domain Tracking spreadsheet [Appendix A]. In addition, under Pathophysiological manifestations/abnormalities, the investigators have identified if this is a Symptom, a Sign, or a Biomarker (imaging, blood work). In total there are 25 domains being considered for inclusion in the REDCap.

The Domain Tracking spreadsheet will be reviewed for completeness by the OMERACT and used as the resource for domains to be entered into REDCap once the protocol has been completed and approved.

Consensus Criteria for e-DelphiSurvey Consensus agreement is defined by over 70% of both stakeholder groups (Patient Research Partners vs Other Stakeholders) voting that the domain is critically important to include (scoring 7 to 9 on the 1 to 9 scale) or not important to include in the Core Domain Set being developed (scoring 1 to 3) over a minimum of two rounds of e-Delphi. Once a domain has reached this level on two rounds, it will be considered as having reached consensus for inclusion or exclusion. Consensus by one group but not both groups will be considered important, but not full consensus. These domains may be worth inclusion as optional domains, or ones requiring further research and discussion. Domains that reach consensus levels in Rounds 1 and 2 (for either inclusion or exclusion) will not be presented in Round 3 for voting, however, they will be presented as the list of domains where consensus had been reached.

Sample Size Oversampling will be done at baseline to allow for attrition of 50%. Since the investigators aim to have a response from 200 patients and 200 other stakeholder members by the end of the final round, the investigators will recruit 800 participants (400 in each group).

Methods Conducting the e-Delphi Survey Initial Soliciting Email and Registration

When the survey is ready and activated, invitees will receive an email and be directed to the survey site for registration. Participants will be asked to enter their age, gender, race, education, income and country of residence. It will also contain a stakeholder group determination field. Depending if the study participant is a patient or physician, the following additional information will be collected on the registration page:

* Years of clinical practice (physician participants only)
* Area of specialization (physician participants only)
* Number of SLE patients accessed per year (physician participants only)
* SLE disease duration (patient participants only)
* Status of SLE treatment (patient participants only)

Once registration is completed, the system will automatically generate Study ID that will be sent to the participant for login of future rounds. At that point they will be directed to the survey for round 1.

The participant's email address and study ID will be used in the REDCap system for linking respondents to their previous responses when they move to subsequent rounds of e-Delphi survey and for email reminders about the survey.

Rounds Three rounds and a 4th sorting round. The first three rounds are an e-Delphi Survey for rating the importance of the domains for inclusion in the Core Domain Set in this area. Core domains are clearly defined as those minimal set of domains (usually numbering 7 or less) that are measured in all clinical trials or research in the defined field. Respondents will be asked to rate the importance of each domain for consideration in the development of this Core Domain Set on a scale of 1-9.

Comment fields are available after each domain to allow people to add additional notes about their decision. At the end of the list of domains there will be a chance for the respondents to nominate additional domains that they felt were missed.

Round 1 will be opened and continue until the sample size is achieved in each stakeholder group (Patients, Others). Results of Round 1 are returned to the working group for consideration of response, new items, and comments. The working group will work between round 1 and 2 to review all recommended domains and will track decisions for inclusion and exclusion; this spreadsheet will include the list of items added and comments on items where there is agreement & disagreement. Domain labels or definitions can be revised to clarify based on these comments. Modifications and additions are made to the REDCap, and the results are advanced for Round 2.

In Round 2 all domains will again be offered along with any newly nominated domains from Round 1. All domains will again be rated for their importance for inclusion. In this situation, the respondents will see their own responses from Round 1 highlighted, and the responses from the other stakeholder groups displayed. The working group will determine a schedule for system reminders and send reminders to Round 1 participants. Groups will work to maintain participant engagement considering the final desired sample size. Round 2 results will be compiled by the software and any domain that has reached consensus for inclusion will move to round 3.

In Round 3, the shorter list of domains that are still yet at the point of consensus are re-evaluated by participants.

Final round A final round gathers all domains that had reached consensus to include in a core domain set for final comment. In this final round, the respondents will be able to select up to 10 domains and upon selection of their choice, they will be asked to offer comments on saying why this domain should or should not, in their opinion, be included. Domains where consensus was to exclude, or those where there is no consensus (no group voting > 70% to include or to exclude) will not be offered in the final round.

This feedback along with the results of all three rounds of the e-Delphi process will be provided to the Working Group in a de-identified format on an Excel spreadsheet to the working group who will use the results and the comments to make their final evidence-based decisions on the content of each layer of the OMERACT Onion, resulting in a OMERACT Core Domain Set.

Management of Non or Partial Responders After implementing the reminder strategies above any non-responders from previous rounds will be excluded from subsequent rounds. Partial responders will be identified in the data and will be excluded from subsequent rounds.

Data Analysis Each round of the Delphi will have a separate analysis of data. Responses from the first round will be summed providing a ranking for each domain based on their Likert scale scores for all respondents, patients only, and other collaborators only. Additionally, the OMERACT SLE Steering Committee will review the suggested domains from all participants and will discuss and decide if any suggested domains should be included in future rounds. Respondents will be provided with their response and the group average in the 2nd round.

Data from the second round will again be summed scores for all respondents, patients only, and other collaborators only. Domains which meet the inclusion or exclusion criteria will be removed from future rounds of the Delphi. Respondents will be provided with their response from round 2 compared to the patient group and other collaborator group separately in the 3rd round.

Data from the third round of the survey will again be summed scores for all respondents, patients only, and other collaborators only. Domains which meet the inclusion or exclusion criteria will be removed from proceeding to the 4th round of the Delphi. Respondents will be provided with their response from round 4 compared to the patient group and other collaborator group separately in the 4th round.

Written responses in round 4 will be reviewed by the OMERACT SLE Steering Committee. The scores for domains when they were removed for inclusion or exclusion or their final scores from the 3rd round along with the comments from the 4th round will be considered as the endpoint scores/comments for each domains. The OMERACT SLE Steering Committee will use these values/comments to organize domains by importance. The range/concentration of participant scores (looking at standard deviation) as well as the mean will be used to prioritize domains, which will be influenced by the judgement of the OMERACT SLE Steering Committee on the comments on domains from the 4th round.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females
2. 18 and older
3. Able to read and understand English, Spanish, French, Italian, Portuguese, Japanese, Arabic, Korean, Hebrew, German, and Chinese
4. Have access to email and the internet

Exclusion Criteria:

1. Not able to read and understand English, Spanish, French, Italian, Portuguese, Japanese, Arabic, Korean, Hebrew, German, and Chinese
2. Does not have access to email and the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: As part of developing and implementing a Core Outcome Set engagement of various stakeholders is essential. The working group will work to engage various stakeholders using the framework below as well as representation from a minimum of 3 continents. 200 SLE patients and 200 other stakeholders will be approached for recruitment. Stakeholder groups include:
  Patients/Public: Individuals receiving or advocating for patient-centered care. Providers: Healthcare professionals and organizations delivering care. Purchasers: Entities underwriting healthcare costs (e.g., employers, governments).
  Payers: Those reimbursing care (e.g., insurers, Medicare). Policy Makers: Regulatory and legislative bodies (e.g., FDA, HHS). Product Makers: Drug and device manufacturers. Researchers: Principal investigators and their funders.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
SLE Core Domain Set as determined by a 4-round Delphi survey | 6 months
  A 4-round Delphi survey will be conducted to ascertain preliminary opinions on the importance of domains measured in SLE to develop a Core Domain Set.
  Once all 4 rounds of the Delphi are complete the feedback along with the results of all three rounds of the Delphi process will be provided to the Working Group in an anonymous format who will use the data of the voting rounds, the selection of the most important domains, and the comments to make their final evidence-based decisions on the content of Core Domain Set. The draft Core Domain Set will be presented the OMERACT Community for endorsement.

CONTACTS AND LOCATIONS:
Overall Officials: Zahi Touma, MD, PhD, Principal Investigator — University Health Network and University of Toronto

IPD SHARING:
Plan to Share IPD: No